CLINICAL TRIAL: NCT04674553
Title: Effect of Obesity Among COVID-19 Patients in Critical Care Settings
Status: Completed | Type: Observational
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Mehwish Iftikhar, Principal Inevstigator, Services Institute of Medical Sciences, Pakistan
Other Study IDs: 16021982
Record Dates: First submitted 2020-12-16; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Obesity; Covid19
Keywords: obesity covid-19 assisted ventilation
MeSH Terms: conditions — Obesity; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A novel human coronavirus that is now named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) (formerly called HCoV-19) emerged in Wuhan, China, in late 2019 and is now causing a pandemic. Human-to-human transmission is primarily achieved through close contact of respiratory droplets, direct contact with the infected individuals, or by contact with contaminated objects and surfaces. As a new chapter in human life opens up, the world seems to be divided into two parts pre- and post-COVID-19 era. Body mass index (BMI) is widely used to define obesity and overweight in adults. A BMI between 25 and 30 indicates overweight and above 30 indicates obesity. It is important to note that the levels of the inflammatory cytokines found in obese people are significantly higher than those in lean people, but they are still lower than those in individuals with infection or trauma. Obesity-mediated alterations in the airways and immune system are extremely important at the present moment considering SARS-Cov-2 infection. This study is designed to determine the effect of overweight and obesity with outcomes of patients with moderate to severe COVID-19 infection in critical care setting. Also, to see outcomes of assisted ventilation in obese patients.

This may help in establishing strong association of obesity with COVID-19 in our part of the world. This may open new treatment strategies for COVID-19 by treating obesity as an essential risk factor.

DETAILED DESCRIPTION:
This Prospective Cohort Study study will be conducted in COVID-19 Intensive care unit, Services hospital Lahore. it will be completed in 3 months after approval of proposal taking 100 patients using Non Probability Purposive sampling.

After ethical approval, research will be started and patients will be recruited from ICU according to inclusion and exclusion criteria. Patients will be randomized to two groups Group A with normal BMI and Group B having over weight and obese patients. They will be given standard treatment as practiced and outcome will be measured in terms of recovery from disease or death. Duration of stay in hospital, progression of disease, O2 requirement, improvement in biochemical profile and radiology or occurrence of complications.

Data will be put in SPSS version 25 and analysis will be done.

ELIGIBILITY:
Inclusion Criteria:

1. All Patients presented to ICU with PCR positive for Covid-19 .
2. Both genders included.
3. Age range 18 to 80 years.
4. Patients fulfilling Criteria for moderate to severe disease.
5. Conscious patient on initial presentation.
6. BMI range from 18-> 40.

Exclusion Criteria:

1. Unable to provide free informed consent.
2. Pregnant females.
3. Gross ascites, amputation or other conditions making BMI measurement unreliable.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Asian people having COVID-19 PCR positive
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | From date of randomization until the date of death from any cause assessed up to 4weeks of study
  COVID-19 related mortality
Recovery from COVID-19 | From date of randomization until recovery and discharge from hospital assessed up to 4weeks of study
  Negative PCR for COVID-19 and discharge from hospital

SECONDARY OUTCOMES:
COVID-19 severity | From date of randomization until the date of first documented symptom progression assessed up to 4weeks of study
  Mild: Asymptomatic; Moderate:; Severe:; Critical: Any one of ARDS or MOF or septic shock
Oxygen requirement | From date of randomization until date of first documented progression assessed up to 4weeks of study
  Mild:SpO2 >94%; Moderate: SpO2<94%; Severe: SpO2<90% but > 80%; Critical: SpO2<80%

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Iftikhar, FCPS (Endo), Principal Investigator — SIMS
Locations (1):
- Mehwish Iftikhar, Lahore, Punjab Province, Pakistan